CLINICAL TRIAL: NCT04724317
Title: Ultrasound Guided Shoulder Intra-Articular Ozone Injection Versus Pulsed Radiofrequency Application for Shoulder Adhesive Capsulitis - A Randomized Controlled Clinical Study
Brief Title: Ultrasound Guided Shoulder Intra-Articular Ozone Injection Versus Pulsed Radiofrequency Application for Shoulder Adhesive Capsulitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ahmed Foula (Other)
Responsible Party: Sponsor-Investigator, Ahmed Foula, Principal Investigator, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1216-4-010
Record Dates: First submitted 2021-01-16; First posted 2021-01-26 (Actual); Last update posted 2022-07-08 (Actual); Status verified 2022-07

CONDITIONS: Adhesive Capsulitis; Shoulder Pain
Keywords: adhesive capsulitis; soulder pain; triamcinolone; ozone; pulsed radiofrequency
MeSH Terms: conditions — Bursitis; Shoulder Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Steroid Group (Sham Comparator): shoulder intra-articular injection of 5 ml of Bupivacaine 0.125% added to triamcinolone 40 mg under the ultrasound guidance
  Interventions: Procedure: Steroid Group
- Ozone Group (Active Comparator): shoulder intra-articular injection of 5 ml of Bupivacaine 0.125% followed by injection of 10 ml of Oxygen-Ozone mixture (15 µg/ml) under the ultrasound guidance
  Interventions: Procedure: Ozone Group
- PRF Group (Active Comparator): shoulder intra-articular injection of 5 ml of Bupivacaine 0.125% followed by pulsed radiofrequency application under the ultrasound guidance
  Interventions: Procedure: PRF Group

INTERVENTIONS:
Procedure: Steroid Group — Ultrasound guided shoulder intra-articular steroid injection
  Arms: Steroid Group
Procedure: Ozone Group — Ultrasound guided shoulder intra-articular Ozone injection
  Arms: Ozone Group
Procedure: PRF Group — Ultrasound guided shoulder intra-articular pulsed radiofrequency application
  Arms: PRF Group

SUMMARY:
The aim of this study is to evaluate the efficacy of the ultrasound guided shoulder intra-articular Ozone injection versus pulsed radiofrequency application in patients with shoulder adhesive capsulitis.

* Primary Outcome :

  - Pain score using visual analogue scale during rest (VASr) and movement (VASm).
* Secondary Outcome :

  * Quality of life using Shoulder Pain and Disability Index (SPADI). It assesses the overall functionality of the shoulder joint.
  * Levels of serum ICAM -1, and serum high sensitive C-reactive protein (hs-CRP) are compared before and after treatment intervention.

DETAILED DESCRIPTION:
After approval of the local ethical committee of Medical Research Institute - Alexandria University (IORG0008812), an informed written consent will be taken from all patients participating in the study. The study will be carried out on 45 adult patients (15 per group) of either gender, aged from 30 to 65 years. Eligible patients are those who were diagnosed with primary shoulder adhesive capsulitis according to the previously mentioned diagnostic criteria, with history of inadequate response to a trial of conservative therapy (NSAIDs and physiotherapy) for at least four weeks.

Patients will be assigned into three equal groups using computerized random blocks method:

1. Steroid Group (S): [15 patients] Control group treated with intra-articular injection of 5 ml of Bupivacaine 0.125% added to triamcinolone 40 mg under the ultrasound guidance.
2. Ozone Group (O3): [15 patients] Patients will be treated with intra-articular injection of 5 ml of Bupivacaine 0.125% followed by injection of 10 ml of Oxygen-Ozone mixture (15 μg/ml) under the ultrasound guidance.
3. Pulsed radiofrequency Group (PRF): [15 patients] Patients will be treated with shoulder intra-articular injection of 5 ml of Bupivacaine 0.125% followed by pulsed radiofrequency application under the ultrasound guidance.

Patients' Evaluation and Preparation:

Patients' preparation starts with pre-intervention evaluation visit. Proper history taking and clinical examination will be carried out. Documentation of the range of motion and VAS score will be done after proper explanation. Patients will be asked to fill a SPADI score form.

Laboratory investigations will include complete blood count (CBC), prothrombin time (PT), and international normalized ratio (INR).

Baseline serum ICAM-1 level and hs-CRP level will be measured using 5 ml of patient's venous blood.

Patients will be asked to sign a consent form to participate in the study. Participants will be admitted to pain management ward. Random assignment will be carried out using computerized random blocks with variable block size.

All interventions will be carried out in the operating theatre (OR) for proper monitoring and sterilization procedures. A 20 G intravenous (IV) cannula will be inserted for all patients in the OR. Basic monitoring will be applied; continuous electrocardiogram (ECG) monitoring, arterial Oxygen saturation (SPO2) monitoring, and non-invasive blood pressure (NIBP) monitoring.

Intervention Methodology:

1. Group S:

   Patients will be put in lateral semi-prone position with the affected shoulder facing up. Shoulder space will be opened by arm internal rotation and adduction across the chest. Under sterile conditions and proper draping of the affected shoulder, scanning will start using Sonosite® M- turbo™ ultrasound machine. A high frequency linear probe (7-14 MHz) will be put parallel and just inferior to spine of the scapula. Identification of humeral head, joint capsule, labrum, glenoid, and infraspinatus and deltoid muscles should be available in one image to avoid wrong needle positioning. The in-plane posterior approach for intra-articular injection will be used (Furman et al., 2017). Needle insertion (22 Gauge, 5 cm length) approach from inferomedial to superolateral direction towards the humeral head. The targeted needle path should avoid labrum puncture. The end point for injection is subcapsular and adjacent to the labrum.

   After confirmation of proper needle position, 5 ml of Bupivacaine 0.125% will be injected added to triamcinolone 40 mg (Babaei-Ghazani et al., 2019).
2. Group O3:

   Under the previously described position and scanning technique, intra-articular injection of 5 ml of Bupivacaine 0.125% followed by 10 ml of Oxygen-Ozone mixture (15 μg/ml) will be done (Noori-Zadeh et al., 2019).
3. Group PRF:

Under the previously described position and scanning technique, 5 ml of Bupivacaine 0.125% will be directly injected. Following, Intra-articular PRF will be applied with a 10 cm neurotherm needle with 10 mm active tip for 4 minutes to the glenohumeral joint (Ozyuvaci et al., 2011).

Post-Procedure Assessment:

All participants will be treated as day-case patients and will be observed in the recovery ward for 2 h after therapy. VAS, shoulder joint ROM, and any complication (e.g., hematoma formation, vasovagal attack, etc.) will be recorded before discharge.

Follow-up visits will be planned for all participants at week 1, 2, 4, 8 post-intervention. During these visits, reassessment will be done for VASr, VASm, SPADI score, and ROM.

* Pain score Using visual analogue scale during rest (VASr) and movement (VASm), pain will be categorized as mild (0-3), moderate (4-6), or severe (7-10). Improved pain score is considered significant when there is a categorical improvement in pain level.
* Quality of life Using Shoulder Pain and Disability Index (SPADI), improvement in quality of life is considered significant when there is 10% reduction in the final index.

During the last follow-up visit, samples for serum ICAM-1 and highly sensitive CRP levels will be obtained.

Statistical Analysis:

Data will be analyzed using descriptive statistical methods as well as comparison of the qualitative and quantitative data. Presentation will be carried out in the form of proper tables and graphical presentation.

ELIGIBILITY:
Inclusion Criteria:

* Aged from 30 to 65 years
* Either gender
* Diagnosed with Adhesive Capsulitis
* Inadequate response for conservative therapy (NSAIDs and physiotherapy) for four weeks

Exclusion Criteria:

* Patients diagnosed with central post-stroke neuropathic pain
* Patients with documented rheumatoid arthritis
* Patients with current shoulder fracture or trauma
* Known causes for secondary adhesive capsulitis (e.g., diabetes)
* Patients with local tumor at shoulder region
* Patients with local skin infection over shoulder region
* Patients with reported coagulopathy
* Patients with allergy to LA

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2021-01-05 (Actual); Primary Completion 2022-06-10 (Actual); Study Completion 2022-06-10 (Actual)

PRIMARY OUTCOMES:
Pain score, using Visual Analogue Scale (VAS) | Initial assessment visit + Immediate post-intervention + Follow-up visits will be planned at week 1, 2, 4, 8 post-intervention.
  Visual analogue scale during rest (VASr) and movement (VASm), pain will be categorized as mild (0-3), moderate (4-6), or severe (7-10). Change in pain score is considered significant when there is a categorical shift in pain level.

SECONDARY OUTCOMES:
QOL improvement, using Shoulder Pain And Disability Index (SPADI) | Initial assessment visit + Immediate post-intervention + Follow-up visits will be planned at week 1, 2, 4, 8 post-intervention.
  Assesses the overall functionality of the shoulder joint. Using SPADI score, change in QOL is considered significant when there is 10% change in the final index.
Systemic inflammatory markers, using serum Intracellular Adhesion Molecule (ICAM 1) level. | Immediate pre-intervention (baseline) + 8 weeks post-intervention (last follow-up visit).
  Levels of serum ICAM -1 are compared before intervention and at the end of follow-up period.
Systemic inflammatory markers, using serum High Sensitive C Reactive Protein (hs-CRP) level. | Immediate pre-intervention (baseline) + 8 weeks post-intervention (last follow-up visit).
  Levels of serum high sensitive C Reactive Protein (hs-CRP) are compared before intervention and at the end of follow-up period.

CONTACTS AND LOCATIONS:
Overall Officials: Laila S. Sabry, MD, Study Director — Department of Anaesthesia and Pain Medicine - Medical Research Institute - Alexandria University; Ahmed F. Elmulla, MD, Study Director — Department of Anaesthesia and Pain Medicine - Medical Research Institute - Alexandria University; Maher A. Kamel, MD, Study Director — Department of Biochemistry - Medical Research Institute - Alexandria University; Adel I. Hozein, MD, Study Director — Department of Anaesthesia and Pain Medicine - Medical Research Institute - Alexandria University
Locations (1):
- Medical Research Institute - Alexandria University, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Yes
All IPD collected can be shared with other researchers in other studies as decided by the main investigator. Personal data will never be shared.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available once be collected and reported in study database.
Access Criteria: All IPD collected can be shared with other researchers in other studies as decided by the main investigator. Personal data will never be shared.

REFERENCES:
- [Background] Angst F, Schwyzer HK, Aeschlimann A, Simmen BR, Goldhahn J. Measures of adult shoulder function: Disabilities of the Arm, Shoulder, and Hand Questionnaire (DASH) and its short version (QuickDASH), Shoulder Pain and Disability Index (SPADI), American Shoulder and Elbow Surgeons (ASES) Society standardized shoulder assessment form, Constant (Murley) Score (CS), Simple Shoulder Test (SST), Oxford Shoulder Score (OSS), Shoulder Disability Questionnaire (SDQ), and Western Ontario Shoulder Instability Index (WOSI). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11:S174-88. doi: 10.1002/acr.20630. No abstract available. PMID 22588743
- [Background] Babaei-Ghazani A, Fadavi HR, Eftekharsadat B, Ebadi S, Ahadi T, Ghazaei F, Khabbaz MS. A Randomized Control Trial of Comparing Ultrasound-Guided Ozone (O2-O3) vs Corticosteroid Injection in Patients With Shoulder Impingement. Am J Phys Med Rehabil. 2019 Nov;98(11):1018-1025. doi: 10.1097/PHM.0000000000001240. PMID 31188145
- [Background] Bak K, Isaksson F. [Frozen shoulder]. Ugeskr Laeger. 2019 Feb 11;181(7):V03180207. Danish. PMID 30777592
- [Background] Basta M, Sanganeria T, Varacallo MA. Anatomy, Shoulder and Upper Limb, Suprascapular Nerve. 2022 Oct 3. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK557880/ PMID 32491803
- [Background] Binder AI, Bulgen DY, Hazleman BL, Roberts S. Frozen shoulder: a long-term prospective study. Ann Rheum Dis. 1984 Jun;43(3):361-4. doi: 10.1136/ard.43.3.361. PMID 6742896
- [Background] Chang LR, Anand P, Varacallo MA. Anatomy, Shoulder and Upper Limb, Glenohumeral Joint. 2025 Mar 3. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK537018/ PMID 30725703
- [Background] Franz A, Klose M, Beitzel K. [Conservative treatment of frozen shoulder]. Unfallchirurg. 2019 Dec;122(12):934-940. doi: 10.1007/s00113-019-00731-3. German. PMID 31650192
- [Background] Kim YS, Kim JM, Lee YG, Hong OK, Kwon HS, Ji JH. Intercellular adhesion molecule-1 (ICAM-1, CD54) is increased in adhesive capsulitis. J Bone Joint Surg Am. 2013 Feb 20;95(4):e181-8. doi: 10.2106/JBJS.K.00525. PMID 23426775
- [Background] Lipov EG, Navaie M, Rothfeld C, Kelzenberg B, Sharghi LH, Solomon DJ, Provencher MT. Use of intra-articular and intrabursal pulsed radiofrequency for the treatment of persistent arthrogenic shoulder pain. Pain Med. 2013 Apr;14(4):554-6. doi: 10.1111/pme.12073. Epub 2013 Mar 14. No abstract available. PMID 23489372
- [Background] Neviaser AS, Neviaser RJ. Adhesive capsulitis of the shoulder. J Am Acad Orthop Surg. 2011 Sep;19(9):536-42. doi: 10.5435/00124635-201109000-00004. PMID 21885699
- [Background] Noori-Zadeh A, Bakhtiyari S, Khooz R, Haghani K, Darabi S. Intra-articular ozone therapy efficiently attenuates pain in knee osteoarthritic subjects: A systematic review and meta-analysis. Complement Ther Med. 2019 Feb;42:240-247. doi: 10.1016/j.ctim.2018.11.023. Epub 2018 Nov 28. PMID 30670248
- [Background] Ozyuvaci E, Akyol O, Acikgoz A, Leblebici H. Intraarticular pulsed mode radiofrequency lesioning of glenohumeral joint in chronic shoulder pain: 3 cases. Korean J Pain. 2011 Dec;24(4):239-41. doi: 10.3344/kjp.2011.24.4.239. Epub 2011 Nov 30. No abstract available. PMID 22220248
- [Background] Su YD, Lee TC, Lin YC, Chen SK. Arthroscopic release for frozen shoulder: Does the timing of intervention and diabetes affect outcome? PLoS One. 2019 Nov 11;14(11):e0224986. doi: 10.1371/journal.pone.0224986. eCollection 2019. PMID 31710642
- [Background] Boonstra AM, Schiphorst Preuper HR, Reneman MF, Posthumus JB, Stewart RE. Reliability and validity of the visual analogue scale for disability in patients with chronic musculoskeletal pain. Int J Rehabil Res. 2008 Jun;31(2):165-9. doi: 10.1097/MRR.0b013e3282fc0f93. PMID 18467932
- [Background] Charan J, Biswas T. How to calculate sample size for different study designs in medical research? Indian J Psychol Med. 2013 Apr;35(2):121-6. doi: 10.4103/0253-7176.116232. PMID 24049221
- [Background] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343
- [Background] Kingston K, Curry EJ, Galvin JW, Li X. Shoulder adhesive capsulitis: epidemiology and predictors of surgery. J Shoulder Elbow Surg. 2018 Aug;27(8):1437-1443. doi: 10.1016/j.jse.2018.04.004. Epub 2018 May 25. PMID 29807717
- [Background] Pannucci CJ, Wilkins EG. Identifying and avoiding bias in research. Plast Reconstr Surg. 2010 Aug;126(2):619-625. doi: 10.1097/PRS.0b013e3181de24bc. PMID 20679844
- See also: Atlas of Image-Guided Spinal Procedures E-Book — https://books.google.com.eg/books?id=e4o-DwAAQBAJ